CLINICAL TRIAL: NCT01794130
Title: The Incidence of Subclinical High-altitude Pulmonary Oedema at High Altitude
Status: Completed | Type: Observational
Sponsor: Institute of Mountain Emergency Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: V/4/11
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Last update posted 2013-02-18 (Estimated); Status verified 2013-02

CONDITIONS: Acute Mountain Sickness; Subclinical High Altitude Pulmonary Edema
MeSH Terms: conditions — Altitude Sickness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this investigation is to determine the incidence of silent interstitial pulmonary edema by chest ultrasound at moderate altitude (3905m). Secondary endpoints are to detect a suspected association with acute mountain sickness (AMS), co-morbidities and endothelial dysfunction (marker of hypoxia responses, endothelial damage and inflammation).

DETAILED DESCRIPTION:
The high-altitude pulmonary edema (HAPE) is the leading cause of death from high altitude sickness. At moderate altitude (2500-4500m) the incidence (0.2-6%) may be underestimated because only clinical HAPE leads to symptoms and motivates the patient to seek medical advice. Cremona et al. [Cremona et al. Pulmonary extravascular fluid accumulation in recreational climbers: a prospective study. Lancet 2002;359:303-09] suggested that a silent interstitial pulmonary edema arises in most recreational climbers at moderate altitude. Recently, chest sonography has been shown to effectively detect pulmonary edema and quantify extravascular lung water through the sign of "ultrasound lung comets" (ULCs) originating from water-thickened interlobular septa [Lichtenstein D et al. The comet-tail artifact. An ultrasound sign of alveolar-interstitial syndrome. Am J Respir Crit Care Med;156:1640-46]. The technique requires only basic twodimensional technology and has been applied in extreme, out-of-hospital setting, showing in recreational climbers a high prevalence of clinically silent interstitial pulmonary edema at high-altitude [Pratali L et al. Frequent subclinical high-altitude pulmonary edema detected by chest sonography as ultrasound lung comets in recreational climbers. Crit Care Med 2010;38:1818-23]. However, data for moderate altitude remain scarce, despite that mountaineers are increasing in age and comorbidities and could be more prone to high altitude emergencies.

Prospective, non-randomised, observational study. Study participants are recruited from a scientific research group lead by the Ohio State University during a glaciology study on the Ortles Glacier in South Tyrol (3905m).

Patients are tested for a baseline measure, during a permanent stay on the glacier camp (3h, 9h, 24h, 48h, 72h, 7d ). Parameters include chest ultrasound, Lake Louise score, cerebral sensitive score, non-invasive haemodynamic parameters (i.e. US) and markers of hypoxia responses, endothelial damage and inflammation.

ELIGIBILITY:
Inclusion Criteria:

* healthy of age >18y

Exclusion Criteria:

* cardiac failure
* chronic kidney disease
* chronic pulmonary disease
* acute lung/heart/kidney/brain conditions
* neoplastic disease
* lack of consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Changes in the number of beta-lines in chest sonography | at 0 (arrival at 3830m), 9, 24, 48 and 72 hours, and at day 7
  as marker of subclinical pulmonary edema

SECONDARY OUTCOMES:
Changes from baseline of optic nerve sheath diameter | at 0 (arrival at 3830m), 3, 9, 24, 48 and 72 hours, and at day 7
  evaluated by optical nerve sonography
Changes from baseline in RNA expression in circulating polymorphonucleated | at 9, 24, 72 hours and day 7

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Strapazzon, MD, Study Director — Institute of Mountain Emergency Medicine, Eurac research
Locations (1):
- Institute of Mountain Emergency Medicine, Eurac research, Bolzano, Provincia autonoma di Bolzano, Italy